CLINICAL TRIAL: NCT02471066
Title: Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on Functional Psychogenic Movement Disorders Followed by a Feasibility Study of a Hypnotherapy Treatment as Adjuvant Therapy.
Brief Title: rTMS Effect in Functional Psychogenic Movement Disorders Applied Alone Then Combined With Hypnotherapy
Acronym: MOVHYSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14 7311 02
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active rTMS (Experimental): 12 patients will be enrolled in this arm.
  Interventions: Device: rTMS
- sham rTMS (Sham Comparator): 12 patients will be enrolled in this arm.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — * Study 1 : 5 daily sessions of rTMS 1 Hz, 95% x resting motor threshold (RMT) applied on M1 / sham
  * Study 2 : 3 weekly sessions of rTMS 1 Hz, 95% x RMT on M1 combined with ericksonian hypnosis session

SUMMARY:
The management of functional psychogenic movement disorders (FNPMD) is challenging for neurologists and psychiatrists and only comprehensive multidisciplinary treatment programme can be worthwhile for these patients (Moene et al 2002). Recent functional magnetic resonance imaging studies have demonstrated abnormalities in motor control at cortical level, hyperactivity of limbic system and disturbance of connectivity between these two systems leading to a lack of self-agency, (Voon et al 2010,2011).Two recent studies suggested a possible therapeutic effect of transcranial magnetic stimulation (TMS) in FNPMD (Dakotakis 2011, Garcin, 2013).

In this protocol our objectives are twofold :

1. to compare the effect of 5 consecutive daily sessions of rTMS on FNPMD in a double-blind randomized controlled study
2. to study the effect of 3 weekly hypnosis sessions combined with rTMS in FNPMD

ELIGIBILITY:
Inclusion criteria:

* Man or woman with FNPMD for at least 2 months,
* diagnosed from clinical Diagnostic and Statistical Manual V conversive somatoform troubles and Gupta & Lang (2009) and Edwards & Bahtia 2012 neurological clinical criteria

Exclusion criteria:

* Severe progressive psychiatric disorders
* Cardiac pace-maker
* Metallic prosthesis
* Cochlear implants
* Previous neurosurgery
* Epilepsy
* Severe cardiac disease
* Alcohol or toxic abuse for the last 12 months
* Drugs such clozapine, bupropion, methadone or theophylline

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changes of Psychogenic Movement Disorder Rating Scale (PMDRS= Hinson score between baseline and one month after rTMS treatment | Inclusion and 1 month later

SECONDARY OUTCOMES:
Clinical Global Impression-Severity scale (CGI-SEVERITY/CGI-I/CGI-S) | inclusion, inclusion + 5 days, inclusion + 1 month, inclusion + 2 months, inclusion + 6 months, inclusion + 12 months.
Hospital Anxiety and Depression Scale (HAD/HDRS) | inclusion, inclusion + 1 month, inclusion + 6 months, inclusion + 12 months.
Quality of Life (SF-36) | inclusion, inclusion + 1 month, inclusion + 2 months, inclusion + 6 months, inclusion + 12 months.
Temperament and Character Inventory (TCI) | inclusion, inclusion + 12 months.
Pain scale (VAS) | : inclusion, inclusion + 5 days, inclusion + 1 month, inclusion + 2 months, inclusion + 6 months, inclusion + 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Toulouse University Hospital, Toulouse, France

REFERENCES:
- [Background] Dafotakis M, Ameli M, Vitinius F, Weber R, Albus C, Fink GR, Nowak DA. [Transcranial magnetic stimulation for psychogenic tremor - a pilot study]. Fortschr Neurol Psychiatr. 2011 Apr;79(4):226-33. doi: 10.1055/s-0029-1246094. Epub 2011 Apr 8. German. PMID 21480152
- [Background] Garcin B, Roze E, Mesrati F, Cognat E, Fournier E, Vidailhet M, Degos B. Transcranial magnetic stimulation as an efficient treatment for psychogenic movement disorders. J Neurol Neurosurg Psychiatry. 2013 Sep;84(9):1043-6. doi: 10.1136/jnnp-2012-304062. Epub 2013 Feb 5. PMID 23385844
- [Result] Taib S, Ory-Magne F, Brefel-Courbon C, Moreau Y, Thalamas C, Arbus C, Simonetta-Moreau M. Repetitive transcranial magnetic stimulation for functional tremor: A randomized, double-blind, controlled study. Mov Disord. 2019 Aug;34(8):1210-1219. doi: 10.1002/mds.27727. Epub 2019 Jun 10. PMID 31180620